CLINICAL TRIAL: NCT02635633
Title: Continuous Thetaburst Stimulation for the Treatment of Refractory Epilepsy - Safety, Feasibility and Proof-of-concept
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty identifying and including eligible patients
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Principal Investigator, Prof. Dr. Kristl Vonck, Prof. Dr. Boon, University Hospital, Ghent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC/2015/0596
Record Dates: First submitted 2015-08-24; First posted 2015-12-21 (Estimated); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Epilepsies, Partial
Keywords: partial epilepsy; unifocal neocortical; treatment resistant; transcranial magnetic stimulation; thetaburst stimulation
MeSH Terms: conditions — Epilepsies, Partial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- continuous thetaburst stimulation (Experimental): Transcranial magnetic stimulation over the epileptogenic focus using a cTBS stimulation protocol.
  Interventions: Device: continuous thetaburst stimulation

INTERVENTIONS:
Device: continuous thetaburst stimulation — On 4 consecutive days patients receive 5 cTBS trains with a 10min intertrain-interval. One cTBS train consists of 600 pulses delivered in bursts at theta frequency (200ms) during 40s. Each burst comprises 3 pulses at 50Hz. Focal stimulation occurs over the epileptogenic focus (EF), perpendicular to the local gyral geometry, using online neuronavigation. Stimulation intensity is set relative to the resting motor threshold (rMT) determined at baseline (80% rMT). Stimulation intensity is further adjusted to the coil-cortex distance at the EF with the following formula: adjusted MT% (AdjMT) = rMT + 2,7*(DEF-DM1) [DEF = distance over EF; DM1 = distance over M1]. If rMT exceeds the capacity of the stimulator output, stimulation intensity is 100% of maximal stimulator output (MSO).
  Other Names: rTMS; cTBS

SUMMARY:
The purpose of this study is to investigate a novel stimulation protocol of repetitive transcranial magnetic stimulation (rTMS) for the treatment of unifocal neocortical epilepsy, namely continuous thetaburst stimulation (cTBS). As this is a pilot study, the primary endpoint is on safety and tolerability of the treatment. However, information on clinical efficacy and mechanism of action will also be collected.

DETAILED DESCRIPTION:
1. Study design:

   This is an open label prospective pilot trial of continuous thetaburst stimulation (cTBS) in patients with unifocal neocortical epilepsy.

   The study comprises a 13-week period, consisting of 4 weeks baseline seizure frequency assessment, a one-week treatment period with baseline assessments on Monday (T0) and stimulation sessions from Tuesday to Friday (T1-T4), and an 8-week follow-up period with short-term assessments immediately after the final stimulation session on Friday afternoon (T4) and long-term assessments after 2 weeks (FU2) and 8 weeks (FU8).
2. Objectives:

   The primary objective is to assess the feasibility, safety and tolerability of cTBS in refractory epilepsy patients. The secondary objectives are to assess the clinical efficacy and associated mechanism of action of cTBS in unifocal neocortical epilepsy.
3. Rationale:

An open label prospective design allows to make a first estimate on the safety, feasibility and tolerability of cTBS in refractory epilepsy patients. There are currently no reports available of cTBS performed in epilepsy patients. The ultimate aim is to assess clinical efficacy of cTBS with regard to seizure frequency, but a feasibility and safety study is a prerequisite in order to achieve this goal.

ELIGIBILITY:
Inclusion Criteria:

* Refractory unifocal neocortical epilepsy with a well-defined ictal onset zone based on a standardized presurgical evaluation
* ≥ 4 seizures/month, for at least six months
* On a stable drug regimen for at least 2 months
* IQ >70
* Reliable completion of a seizure diary by patient or caretakers
* Therapeutic compliance in the past
* Informed consent signed

Exclusion Criteria:

* Pregnancy, short-term birth wish or childbearing age without adequate birth control
* History of psychogenic non-epileptic seizures
* Intracranial metal hardware (excluding dental filling): surgical clips, shrapnell, electrodes under the stimulation area
* Presence of pacemaker, implantable cardioverter-defibrillator (ICD), permanent medication pumps, cochlear implants or deep brain stimulation (DBS)

Patients with a vagus nerve stimulator are not excluded, provided that adequate distance between the coil and the implanted material can be maintained.

As the short duration of the study will not interfere with an ongoing presurgical evaluation and/or its eventual conclusion, the patients in the course of the evaluation or awaiting surgery are also eligible for inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Seizure induction | Throughout stimulation, 4 days
  Induction of epileptic seizures during or in-between rTMS stimulation trains as a measure of safety

SECONDARY OUTCOMES:
Seizure diary | Throughout the study, lasting 13 weeks
  Self-reported seizure frequency throughout the study as a measure of clinical efficacy.
  Four separate seizure diaries are provided:
  * Baseline period: 4 weeks prior to treatment
  * Treatment week: from monday to friday evening
  * Follow-up part 1: two weeks following the treatment week
  * Follow-up part 2: week 3 to week 8 following treatment Patients note down if the seizure was habitual, atypical or if it was an episode of uncertain etiology (eg. non-epileptic)
Adverse events diary | Throughout the study, lasting 13 weeks
  Description of all experienced adverse event during the study as a measure of safety and tolerability.
Number of interictal epileptiform discharges (IEDs) on hd-EEG | Throughout the study, lasting 13 weeks: baseline (before treatment), following final stimulation session (short-term follow-up), 2 weeks after stimulation and 8 weeks after stimulation (long-term follow-up)
  A 15min hd-EEG is recorded and IEDs are counted during acquisition. Comparison of number of IEDs between the different time points as a measure of clinical efficacy.
Number of interictal epileptiform discharges (IEDs) on normal EEG | Throughout the study, lasting 13 weeks: assessment immediately before and after each treatment session
  Fifteen min EEG with 21 scalp electrodes is recorded immediately before and following each stimulation session. Number of IEDs are counted and compared between pre- and post acquisition as a measure of clinical efficacy.
Cortical resting motor threshold (rMT) | Throughout the study, lasting 13 weeks: baseline (before treatment), following final stimulation session (short-term follow-up), 2 weeks after stimulation and 8 weeks after stimulation (long-term follow-up)
  Cortical resting motor threshold is determined using single-pulse TMS over the primary motor cortex (M1) (ipsilateral to epileptogenic focus). Motor-evoked potential (MEP) is measured over the first dorsal interosseus (FDI) of the contralateral hand. Using a threshold tracking tool (Adaptive PEST) the minimally required stimulation intensity that elicits an MEP of 50 microvolt is determined.
  RMT at different time points throughout the study is compared to assess the effect of the treatment on cortical excitability as a measure of mechanism of action.
TMS-EEG evoked potentials (TEPs) | Throughout the study, lasting 13 weeks: baseline (before treatment), following final stimulation session (short-term follow-up), 2 weeks after stimulation and 8 weeks after stimulation (long-term follow-up)
  TMS-EEG evoked potentials are measured over the epileptogenic focus and the primary motor cortex by performing single-pulse TMS (100 consecutive pulses jittered around an interval of 5s) with continuous EEG acquisition. The EEG is processed in order to obtain quantitative and comparable TEPs measures that reflect cortical excitability.
  These TEP measures obtained at different time points throughout the study are compared to assess the effect of the treatment on cortical excitability as a measure of mechanism of action.
Magnetic resonance imaging (MRI) | Throughout the study, lasting 13 weeks: baseline (before treatment), following final stimulation session (short-term follow-up), 2 weeks after stimulation and 8 weeks after stimulation (long-term follow-up)
  Resting-state functional MRI (rs-fMRI) is acquired at the four main time points of the study to assess the effects of treatment on functional connectivity as a measure of mechanism of action.
High-density EEG (hd-EEG) | Throughout the study, lasting 13 weeks: baseline (before treatment), following final stimulation session (short-term follow-up), 2 weeks after stimulation and 8 weeks after stimulation (long-term follow-up)
  A 128-channel EEG for resting-state EEG acquisition is obtained at the four main time points of the study to assess the effects of treatment on functional connectivity as a measure of mechanism of action.
Change in Montreal Cognitive Assessment score (MoCA) | Throughout the study, lasting 13 weeks: baseline (before treatment), following final stimulation session (short-term follow-up) and 8 weeks after stimulation (long-term follow-up)
  Score ranging from 0 [worst cognitive state] to 30 [best cognitive state], with a score of 26 or higher reflecting normal cognitive function. Cognitive assessment as a measure of safety: comparison at different time points throughout the study using MoCA version 7, 7.2 and 7.3 respectively.
Change in Computerized Visual Searching Task (CVST) | Throughout the study, lasting 13 weeks: baseline (before treatment), following final stimulation session (short-term follow-up), 2 weeks after stimulation and 8 weeks after stimulation (long-term follow-up)
  A 24-figure task assessing mean trial time [the faster the better] and number of errors [the lower the better] Assessment of mental flexibility and information processing as a measure of safety: comparison at different time points throughout the study.
Change in Quality of life in epilepsy-31 (QOLIE-31) | Throughout the study, lasting 13 weeks: baseline (before treatment) and 8 weeks after stimulation (long-term follow-up)
  Questionnaire scoring quality of life (QoL) ranged from 0 [lowest QoL] to 100 [highest QoL] (with associated T-value per score) as a measure of well-being.
Change in Beck depression inventory (BDI-II) | Throughout the study, lasting 13 weeks: baseline (before treatment) and 8 weeks after stimulation (long-term follow-up)
  Questionnaire scoring depression ranged from 0 to 63 as a measure of well-being.
Change in Positive affect negative affect schedule (PANAS) | Throughout the study, lasting 13 weeks: baseline (before treatment) and 8 weeks after stimulation (long-term follow-up)
  Questionnaire scoring affect as a measure of well-being.
Change in State-trait anxiety inventory (STAI) | Throughout the study, lasting 13 weeks: baseline (before treatment) and 8 weeks after stimulation (long-term follow-up)
  Questionnaire scoring anxiety as a state (now) or a trait (more generally) separately, ranged from 20 [less anxious] - 80 [more anxious] as a measure of well-being.
Change in Visual analogue scale (VAS) of general well-being | Throughout the study, lasting 13 weeks: baseline (before treatment) and 8 weeks after stimulation (long-term follow-up)
  Score ranged from 0 [lowest well-being] to 100 [highest well-being] as a measure of well-being.
Change in Visual analogue scale (VAS) of tolerability of the treatment | Throughout the study: after each treatment session and at the end of the study (8 weeks after stimulation)
  Score ranged from 0 [absolutely tolerable] -100 [absolutely intolerable] as a measure of tolerability and feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Kristl Vonck, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Sun W, Mao W, Meng X, Wang D, Qiao L, Tao W, Li L, Jia X, Han C, Fu M, Tong X, Wu X, Wang Y. Low-frequency repetitive transcranial magnetic stimulation for the treatment of refractory partial epilepsy: a controlled clinical study. Epilepsia. 2012 Oct;53(10):1782-9. doi: 10.1111/j.1528-1167.2012.03626.x. Epub 2012 Sep 5. PMID 22950513
- [Background] Fregni F, Otachi PT, Do Valle A, Boggio PS, Thut G, Rigonatti SP, Pascual-Leone A, Valente KD. A randomized clinical trial of repetitive transcranial magnetic stimulation in patients with refractory epilepsy. Ann Neurol. 2006 Oct;60(4):447-55. doi: 10.1002/ana.20950. PMID 17068786
- [Background] Cantello R, Rossi S, Varrasi C, Ulivelli M, Civardi C, Bartalini S, Vatti G, Cincotta M, Borgheresi A, Zaccara G, Quartarone A, Crupi D, Lagana A, Inghilleri M, Giallonardo AT, Berardelli A, Pacifici L, Ferreri F, Tombini M, Gilio F, Quarato P, Conte A, Manganotti P, Bongiovanni LG, Monaco F, Ferrante D, Rossini PM. Slow repetitive TMS for drug-resistant epilepsy: clinical and EEG findings of a placebo-controlled trial. Epilepsia. 2007 Feb;48(2):366-74. doi: 10.1111/j.1528-1167.2006.00938.x. PMID 17295632
- [Background] Theodore WH, Hunter K, Chen R, Vega-Bermudez F, Boroojerdi B, Reeves-Tyer P, Werhahn K, Kelley KR, Cohen L. Transcranial magnetic stimulation for the treatment of seizures: a controlled study. Neurology. 2002 Aug 27;59(4):560-2. doi: 10.1212/wnl.59.4.560. PMID 12196649
- [Background] Nyffeler T, Wurtz P, Luscher HR, Hess CW, Senn W, Pflugshaupt T, von Wartburg R, Luthi M, Muri RM. Repetitive TMS over the human oculomotor cortex: comparison of 1-Hz and theta burst stimulation. Neurosci Lett. 2006 Nov 27;409(1):57-60. doi: 10.1016/j.neulet.2006.09.011. Epub 2006 Oct 17. PMID 17049743
- [Background] Nyffeler T, Cazzoli D, Hess CW, Muri RM. One session of repeated parietal theta burst stimulation trains induces long-lasting improvement of visual neglect. Stroke. 2009 Aug;40(8):2791-6. doi: 10.1161/STROKEAHA.109.552323. Epub 2009 Jun 11. PMID 19520986
- [Background] Goldsworthy MR, Pitcher JB, Ridding MC. The application of spaced theta burst protocols induces long-lasting neuroplastic changes in the human motor cortex. Eur J Neurosci. 2012 Jan;35(1):125-34. doi: 10.1111/j.1460-9568.2011.07924.x. Epub 2011 Nov 25. PMID 22118241
- [Derived] Carrette S, Boon P, Klooster D, Van Dycke A, Carrette E, Miatton M, Raedt R, Delbeke J, Meurs A, Vonck K. Continuous theta burst stimulation for drug-resistant epilepsy. Front Neurosci. 2022 Aug 17;16:885905. doi: 10.3389/fnins.2022.885905. eCollection 2022. PMID 36061598